CLINICAL TRIAL: NCT01313286
Title: The Relative Bioavailability of a Proposed Phase 2 LY2608204 Test Formulation Compared With the Current Phase 1 LY2608204 Reference Formulation After Administration of a Single Oral 80-mg Dose in Healthy Subjects
Brief Title: A Study to Compare Two Forms of LY2608204 in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14233; I3P-FW-GKBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glucokinase activator compound 50

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2608204 Reference, LY2608204 Test (Experimental): Single oral 80 mg dose of LY2608204 reference formulation in period 1; single oral 80 mg dose of LY2608204 test formulation in period 2. There is a washout period of at least 14 days between dosing periods.
  Interventions: Drug: LY2608204 Reference; Drug: LY2608204 Test
- LY2608204 Test, LY2608204 Reference (Experimental): Single oral 80 mg dose of LY2608204 test formulation in period 1; single oral 80 mg dose of LY2608204 reference formulation in period 2. There is a washout period of at least 14 days between dosing periods.
  Interventions: Drug: LY2608204 Reference; Drug: LY2608204 Test

INTERVENTIONS:
Drug: LY2608204 Reference — Administered orally
  Other Names: Glucokinase Activator
Drug: LY2608204 Test — Administered orally.
  Other Names: Glucokinase Activator

SUMMARY:
The purpose of this study is to compare 2 formulations of the study drug (LY2608204) in terms of how much gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy male or a female who cannot become pregnant
* Must have body mass index (BMI) of 18.5 to 32 kg/m², inclusive
* Blood pressure as well as blood and urine laboratory test results must be acceptable for the study
* The veins must be suitable for easy blood collection
* Must be willing to be available for the whole study and be willing to follow study procedures
* Must have given written informed consent

Exclusion Criteria:

* Were in another new drug or medical research study in the last 30 days
* Have participated in this study or any other study with LY2608204 before
* Have taken drugs similar to LY2608204 (glucokinase activators) before and was found to be allergic to the drug
* Have drug allergy to more than 3 types of medications given by injection
* Currently have or used to have health problems or laboratory test results that in the opinion of the doctor, could interfere with understanding the results of this study
* Electrocardiogram (ECG) readings are not suitable for the study
* Are infected with hepatitis B
* Are infected with human immunodeficiency disease virus (HIV)
* Are using or intend to use over-the-counter medication or prescription medications within 14 days, from the start of the first study dosing until end of study
* Are unwilling to follow dietary restrictions/requirements for the study including (i) refrain from consuming foods or beverages containing grapefruit pomelo, star fruit, or Seville orange within 14 days of the start of the study drug dosing until collection of the last blood sample for drug assay; (ii) consume only the meals provided during dosing day at the clinical research unit (CRU)
* Have a regular alcohol intake greater than 21 units per week (males) and 14 units per week (females) or are not willing to abstain from alcohol while in the research unit
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic
* Have a history of drug or alcohol abuse
* Have donated 450 milliliter (mL) or more of blood in the last 3 months (this is about the same as the usual volume given in a blood donation)
* The study doctor thinks the subject should not participate for any other reasons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2608204 Reference, LY2608204 Test: A single oral dose of 80 mg LY2608204 reference formulation in Period 1 and a single oral dose of 80 mg LY2608204 test formulation in Period 2. There is a washout period of at least 14 days between dosing periods.
- LY2608204 Test, LY2608204 Reference: A single oral dose of 80 mg LY2608204 test formulation in Period 1 and a single oral dose of 80 mg LY2608204 reference formulation in Period 2. There is a washout period of at least 14 days between dosing periods.
Period: Period 1
Arm/Group | LY2608204 Reference, LY2608204 Test | LY2608204 Test, LY2608204 Reference
Started | 8 | 8
Completed | 6 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Period 2
Arm/Group | LY2608204 Reference, LY2608204 Test | LY2608204 Test, LY2608204 Reference
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: A single oral dose of 80 mg LY2608204 reference formulation in Period 1 and a single oral dose of 80 mg LY2608204 test formulation in Period 2; or a single oral dose of 80 mg test formulation in Period 1 and a single oral dose of 80 mg reference formulation in Period 2. There is a washout period of at least 14 days between dosing periods.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14
  White | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞])
Description: Area under the concentration versus time curve from zero to infinity [AUC(0-∞)] was calculated from the data. The values for AUC were log-transformed and analyzed using a linear mixed effects model with fixed factor for formulation, sequence and period, and a random factor for subject.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 and 168 hours
Population: All randomized participants who took at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hour per milliliter (ng.h/mL)
Groups:
- LY2608204 Free Base (Reference Formulation): a single oral dose of 80 mg LY2608204 reference formulation (free base)
- LY2608204 Hydrochloride (HCl) Salt (Test Formulation): a single oral dose of 80 mg LY2608204 test formulation (HCl salt)
Arm/Group | LY2608204 Free Base (Reference Formulation) | LY2608204 Hydrochloride (HCl) Salt (Test Formulation)
Number analyzed (Participants) | 16 | 14
nanogram.hour per milliliter (ng.h/mL) | 974 (39) | 1080 (35)
Statistical Analysis 1: Comparison: LY2608204 Free Base (Reference Formulation) vs LY2608204 Hydrochloride (HCl) Salt (Test Formulation); Test type: Superiority or Other; Mixed Models Analysis; Ratio of test formulation (HCl salt) to reference formulation (free base); Ratio of Geometric Least Square means = 1.08, 90% CI 2-sided [1.00 to 1.16]

2. Primary Outcome: Maximum Observed Drug Concentration (Cmax)
Description: Maximum observed drug concentration (Cmax) was observed from the data. The values for Cmax were log-transformed and analyzed using a linear mixed effects model with fixed factor for formulation, sequence and period, and a random factor for subject.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 and 168 hours
Population: All randomized participants who took at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2608204 Free Base (Reference Formulation) | LY2608204 Hydrochloride (HCl) Salt (Test Formulation)
Number analyzed (Participants) | 16 | 14
nanogram per milliliter (ng/mL) | 24.9 (27) | 30.3 (33)
Statistical Analysis 1: Comparison: LY2608204 Free Base (Reference Formulation) vs LY2608204 Hydrochloride (HCl) Salt (Test Formulation); Test type: Superiority or Other; Mixed Models Analysis; Ratio of test formulation (HCl salt) to reference formulation (free base); Ratio of Geometric Least Square means = 1.18, 90% CI 2-sided [1.07 to 1.31]

ADVERSE EVENTS:
Groups:
- LY2608204 Reference Formulation: A single oral dose of 80 mg LY2608204 reference formulation.
- LY2608204 Test Formulation: A single oral dose of 80 mg LY2608204 test formulation.
Arm/Group | LY2608204 Reference Formulation | LY2608204 Test Formulation
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 10/16 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2608204 Reference Formulation (N=16) | LY2608204 Test Formulation (N=14)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 4 (5) | 3 (3)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 4 (5) | 5 (7)
Vessel puncture site reaction (General disorders) | 7 (7) | 2 (2)
Vessel puncture site swelling (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes